CLINICAL TRIAL: NCT03162874
Title: A Multi-centre, Double-blind, Randomised, Placebo-controlled, Parallel-arm Phase IIa Trial to Evaluate the Efficacy, Safety and Tolerability of 28-Day Oral Treatment With PXT002331 (Foliglurax) in Reducing Motor Complications of Levodopa Therapy in Subjects With Parkinson's Disease Experiencing End-of-dose Wearing Off and Levodopa-Induced Dyskinesia (AMBLED)
Brief Title: Study to Evaluate the Efficacy, Safety and Tolerability of PXT002331 (Foliglurax) in Reducing Motor Complications of Levodopa Therapy in Parkinson Disease's Patients
Acronym: AMBLED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prexton Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PXT-CL17-001; 18023A (Other: Lundbeck)
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
Keywords: Levodopa-Induced Dyskinesia (LID); Wearing-off; Foliglurax; Parkinson's Disease; mGluR4 PAM
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PLACEBO (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule
- PXT002331 - 10mg (Experimental)
  Interventions: Drug: PXT002331 - dose 1
- PXT002331 - 30mg (Experimental)
  Interventions: Drug: PXT002331 - dose 2

INTERVENTIONS:
Drug: Placebo oral capsule — BID
  Arms: PLACEBO
Drug: PXT002331 - dose 1 — Oral
  Arms: PXT002331 - 10mg
Drug: PXT002331 - dose 2 — Oral
  Arms: PXT002331 - 30mg

SUMMARY:
This will be a double-blind, randomised, placebo-controlled parallel-arm phase II proof of concept in subjects with PD treated with a stable dose of levodopa who are experiencing both end-of-dose wearing off and Levodopa-Induced Dyskinesia (LID)

ELIGIBILITY:
Inclusion Criteria:

* Males or females diagnosed after the age of 30 years with idiopathic PD for at least 3 years
* Disease severity of 2 to 4 on the modified Hoehn and Yahr scale when in the OFF state
* Been treated with a stable regimen of levodopa-containing therapy
* Subjects who are on a long-acting formulation of levodopa-containing therapy, including Apodespan PR (or equivalent), must be on a stable dose for at least 6 weeks prior to the first screening visit
* Experienced motor fluctuations with wearing off over a period of at least 3 months prior to randomisation
* Experienced LID over a period of at least 3 months prior to randomisation
* Female subjects will be women of non-childbearing potential
* Subjects must pass a Hauser diary concordance test
* Subjects are able, with or without the help of a caregiver, to understand the purpose and risks of the study and provide signed and dated informed consent and authorisation to use confidential health information in accordance with national and local subject privacy regulations

Exclusion Criteria:

* Subjects with atypical, secondary or drug-induced Parkinsonism
* Subjects with a Mini-Mental State Examination (MMSE) score <25
* Any known contraindication to the use of levodopa, including a history of malignant melanoma or a history of narrow-angle glaucoma.
* Subjects who have had a clinically significant illness within 4 weeks of first dose, as determined by the Investigator.
* Any advanced, severe or unstable disease (other than PD) that may interfere with the primary and secondary study outcome evaluations
* Subjects who have undergone prior neurosurgical operation for PD or transcranial magnetic stimulation.
* Subjects who are participating in another clinical study (eg, attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months prior to the baseline visit.
* Female subjects of childbearing potential
* Subjects who are pregnant (as determined by positive serum pregnancy test at screening and/or baseline), breastfeeding or lactating.
* Subjects who, in the opinion of the Investigator, should not participate in this study.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of Treatment Period in the daily awake OFF time based on subject Hauser diary entries | 28 days

CONTACTS AND LOCATIONS:
Locations (45):
- Universitätsklinik für Innere Medizin VI Innsbruck, Neurologisches Studienzentrum, Innsbruck, Austria
- France (14):
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Hôpital Avicenne APHP, Bobigny
  - Hôpital Pierre Wertheimer, Bron
  - CHU Gabriel-Montpied, Clermont-Ferrand
  - CHU Grenoble - Pôle Psychiatrie et Neurologie, Grenoble
  - CHRU - Hôpital Roger Salengro, Lille
  - CHU de Nice - Hôpital Pasteur, Nice
  - Hopital Pitie-Salpetriere, Paris
  - CHU de Poitiers, Poitiers
  - Hôpital Universitaire, Rouen
  - CHU de Nantes - Hôpital Nord Laennec, Saint-Herblain
  - Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hôpital Purpan, Toulouse
- Germany (7):
  - Practice for Neurology, Psychiatry & Psychotherapy Dr. med. I. Schoell & colleagues, Bad Homburg
  - St. Joseph-Krankenhaus Berlin-Weissensee, Berlin
  - University Hospital Erlangen - Abteilung fur Molekulare Neurologie, Erlangen
  - Neurological Praxis, Gera
  - Am Klinikum 1 Jena, Jena
  - Paracelsus-Elena-Klinik Kassel, Kassel
  - MVZ Kliniken Mühldorf a. Inn, Mühldorf
- Italy (11):
  - Villa Margherita, Arcugnano
  - Fondazione Universita G. D'Annunzio Centro Studi sull'invecchiamento Centro di Ricerca Clinica, Chieti
  - Universita degli Studi di Salerno, Fisciano
  - IRCCS Centro Neurolesi Bonino Pulejo, Messina
  - Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento Ospedaliero di Santa Chiara, Pisa
  - Policlinico Tor Vergata, Roma
  - IRCCS San Raffaele Pisana, Roma
  - Università degli Studi di Roma "La Sapienza", Roma
  - Humanitas Research Hospital, Rozzano
  - IRCCS Fondazione Ospedale San Camillo (SC), Venezia
- Spain (7):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (5):
  - Fairfield General Hospital, Bury
  - Imperial College Healthcare NHS Trust - Charing Cross Hospital, London
  - Clinical Ageing Research Unit, Campus for Ageing and Vitality, Newcastle upon Tyne
  - North Tyneside General Hospital, North Shields
  - Plymouth Hospitals NHS Trust - Derriford Hospital, Plymouth